CLINICAL TRIAL: NCT02755168
Title: Feasibility and Outcomes of External Pop-out Versus Classic Fetal Head Extract During Cesarean Section
Brief Title: External Pop-Out Technique Versus Classic Head Extraction During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPO
Record Dates: First submitted 2016-04-23; First posted 2016-04-28 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Caesarean Section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Pop-Out Cesarean Section (Other)
  Interventions: Procedure: External Pop-Out Cesarean Section
- Classic technique (Other)
  Interventions: Procedure: Classic technique

INTERVENTIONS:
Procedure: External Pop-Out Cesarean Section — During fetal head extraction, the obstetrician puts four fingers of his right hand on the lower segment at uterovesical pouch. The palmar aspect of the fingers will be resting on the uterovesical peritoneal reflection not on directly on the fetal head. While the palmar aspect of the fingers was facing the lower segment they were pushed deep below the fetal head.
  Arms: External Pop-Out Cesarean Section
Procedure: Classic technique — During fetal head extraction, the obstetrician puts four fingers of his right hand inside the uterus.
  Arms: Classic technique

SUMMARY:
Caesarean section is one the most common operations worldwide, its rates are globally increasing. A multitude of efforts had been done aiming at reduction of Caesarean section related maternal morbidities; most of them are related to technical modifications of how to open and how to close the abdominal and uterine incisions . The comparative studies of blunt versus sharp extension of the uterine incision showed a reduction of the incidence of unintended extension from 8.8% to 4.8% .

The vulnerability of the lower uterine segment for tears are related to stage of labor. The frequency of unintended extension was reported to be 15.5%, and 35.0% in cases operated in first and second stages of labor respectively.

The original techniques of fetal head extraction entail the introduction of the obstetricians hand or other instruments into the lower uterine segment . This puts the lower uterine segment at risk of damage and incision extensions with its consequences of increased blood loss, increased operative time, infection adhesions and blood transfusion. Adherence to the available the generated good quality evidence bases practice in Caesarean section is anticipated to decease such morbidities.

The idea of the present technique was derived from the fact that during vaginal delivery the main task of obstetrician is to support the perineum while the fetal head extends to get out through birth canal.

ELIGIBILITY:
Inclusion Criteria:

* single fetus
* more than 37 weeks of gestation
* elective Caesarean section

Exclusion Criteria:

* non-cephalic presentation
* placenta previa
* hydrocephalus
* Multiple pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
The success rate of External POP out technique | 20 minutes

SECONDARY OUTCOMES:
Number of women will need blood transfusion | 24 hours
Time of head extraction | 5 minutes
Easiness score: | 5 minutes
  The ES was calculated at a graduated Likert-type scale from zero to 100; in which zero means terribly difficult and 100 means very easy.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided